CLINICAL TRIAL: NCT02412930
Title: Comparative Study of Ultrasound-guided Paravertebral Block Versus Intravenous Tramadol for Postoperative Pain Control in Percutaneous Nephrolithotomy
Brief Title: Comparative Study of Ultrasound-guided Paravertebral Block Versus Intravenous Tramadol in Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra, Assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5/8-2012
Record Dates: First submitted 2015-03-27; First posted 2015-04-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Paravertebral Block (Active Comparator): With ultrasound guidance at T10 to L1 levels, using 0.5% bupivacaine total dose of 15 mL in group P. 5 mL bupivacaine 0.5% was injected in each dermatome level.
  Interventions: Procedure: Ultrasound-guided Paravertebral Block; Drug: Group Tramadol; Drug: Bupivacaine; Device: Ultrasound
- Group tramadol (Placebo Comparator): Patients in group T were given a loading dose of tramadol of 1 mgkg-1
  Interventions: Drug: Group Tramadol

INTERVENTIONS:
Procedure: Ultrasound-guided Paravertebral Block — paravertebral block was performed by ultrasound guidance at T11, T12 and L1 levels, using 0.5% bupivacaine total dose of 15 mL in group P. The injection site was covered with sterile drapes, after cleaning with 10% povidone-iodine solution.
  After, patients in both groups were performed patient controlled analgesia (PCA). The PCA was prepared with 400 mg tramadol into 100 mL of saline. The doses of tramadol in the PCA were bolus dose 0.1 mgkg-1 every 20 minutes without a background infusion.
  Arms: Group Paravertebral Block
Drug: Group Tramadol — Patients in group T were given intravenously a loading dose of tramadol of 1 mgkg-1, 45 minutes before the end of surgery. After,patients in both groups were performed patient controlled analgesia (PCA). The PCA (CADD Legacy PCA pump, Smiths Medical MD, Inc., St. Paul, MN) was prepared with 400 mg tramadol into 100 mL of saline. The doses of tramadol in the PCA were bolus dose 0.1 mgkg-1 every 20 minutes without a background infusion.
Drug: Bupivacaine
  Arms: Group Paravertebral Block
Device: Ultrasound
  Arms: Group Paravertebral Block

SUMMARY:
Paravertebral block has been widely used for analgesia. The aim of this study,comparison of the effect of ultrasound-guided paravertebral block versus intravenous tramadol for postoperative pain control in percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
The study protocol was approved by the Local Ethical Committee. Written informed consent was obtained from all patients, before starting to surgery.

The patients were given no premedication. The demographic data of patients (age, gender, the presence of other diseases) were recorded, preoperatively. All patients were applied standard monitoring in the operating room. After the induction of anesthesia provided intravenously propofol (2-3mg/kg) and rocuronium bromide (0.5 mgkg-1), all patients were intubated with a suitable endotracheal tube. Anesthesia maintenance was provided with 1-2% sevoflurane and a 60% nitrous oxide-40% oxygen gas mixture. 0.9% NaCl (5-10 mLkg-1) was started as fluid resuscitation. Urinary catheter was inserted before placement, and then all patients were placed in the prone position.

Postoperatively, duration of surgery, systolic and diastolic blood pressures, heart rate, peripheral oxygen saturation (SBP, DBP, HR, and SpO2), visual analog scales (VAS), side effects such as vomiting and nausea, complications such as pneumothorax, tramadol consumption and additional analgesic requirements of patients were recorded at 1, 2, 4, 6, 12 and 24 h in the postoperative period. These parameters were evaluated by an anesthesiologist in the first 24 hours postoperatively. If the VAS score was >4, patients in both groups were administered diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* 53 patients scheduled for percutaneous nephrolithotomy (PNL),
* 18-70 years of age,
* weight between 50-100 kg,
* American Society of Anesthesiologists (ASA) classification I-II were included

Exclusion Criteria:

* The exclusion criteria were refusals by patients,
* coagulation abnormalities,
* patients with spinal deformity,
* cutaneous infection at the injection site and
* a known allergy to drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 24 hours
  Postoperative pain degree was evaluated by Visual Analogue Scale

SECONDARY OUTCOMES:
tramadol consumption | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Hatipoğlu, Assist Prof, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

REFERENCES:
- [Derived] Hatipoglu Z, Gulec E, Turktan M, Izol V, Aridogan A, Gunes Y, Ozcengiz D. Comparative study of ultrasound-guided paravertebral block versus intravenous tramadol for postoperative pain control in percutaneous nephrolithotomy. BMC Anesthesiol. 2018 Feb 17;18(1):24. doi: 10.1186/s12871-018-0479-7. PMID 29454333